CLINICAL TRIAL: NCT00993967
Title: A Phase III Open-Label, Single-Group, Extension Study to Obtain Long-Term Safety and Tolerability Data of Idebenone in the Treatment of Friedreich's Ataxia Patients.
Brief Title: Long-Term Safety and Tolerability of Idebenone in Friedreich's Ataxia Patients (MICONOS Extension)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNT-III-001-E
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Results first posted 2018-03-05 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2017-08

CONDITIONS: Freidreich's Ataxia
Keywords: FRDA; idebenone; FRDA disease
MeSH Terms: interventions — idebenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Idebenone (Experimental): 1350 mg/day or 2250 mg/day for patients weighing ≤45 kg or >45 kg, respectively.In case of poor tolerability, dose reduction to 450 mg/day or 900 mg/day, respectively, were allowed.
  Interventions: Drug: idebenone

INTERVENTIONS:
Drug: idebenone — Idebenone 1350 mg/d, patients < or equal 45 kg Idebenone 2250 mg/d, patients > 45 kg

SUMMARY:
This is an Extension study of the MICONOS main randomised placebo-controlled trial (NCT00905268), and open to those patients completing the main study. The scientific aim of this extension study is to monitor safety and tolerability of idebenone over two years in patients with Friedreich's Ataxia.

ELIGIBILITY:
Inclusion Criteria:

* Completion of 52 weeks in study SNT-III-001
* Body weight ≥ 25 kg
* Negative urine pregnancy test
* Eligibility to participate in the present extension study as confirmed by investigator

Exclusion Criteria:

* Safety or tolerability issues arising during the course of SNT-III-001 which in the opinion of the investigator preclude further treatment with idebenone
* Clinically significant abnormalities of haematology or biochemistry including, but not limited to, elevations greater than 1.5 times the upper limit of SGOT, SGPT or creatinine
* Parallel participation in another clinical drug trial
* Pregnancy or breast-feeding
* Abuse of drugs or alcohol

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nick Wood, Professor, Principal Investigator — Dept of Molecular Neuroscience, Institute of Neurology. The National Hospital, University College London
Locations (11):
- Universitätsklinik Innsbruck, Innsbruck, Austria
- Hôpital Erasme - Univeristé Libre de Bruxelles, Brussels, Belgium
- Hôpital de la Salpétrière - INSERM U679, Neurologie et Thérapeutique expérimentale, Paris, France
- Germany (7):
  - HELIOS Klinikum Berlin, Berlin
  - Neurologische Universitätsklinik und Ploklinik - Universitätsklimikum Bonn, Bonn
  - Klinik II, Neuropädiatrie und Muskelerkrankungen - Universitätsklinik Freiburg, Freiburg im Breisgau
  - Zentrum für Neurologische Medizin, Göttingen
  - UKE Hamburg Neuropädiatrie - Zentrum für Frauen, Kinder und Jugendmedizin, Hamburg
  - Neurologische Klinik - Klinikum Grosshadern, München
  - Neurologische Universitätsklinik und Poliklinik, Tübingen
- University medical Center Groningen, Groningen, Netherlands

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Idebenone
Started | 200
Completed | 139
Not Completed | 61
Not completed — Adverse Event | 8
Not completed — Death | 1
Not completed — Lost to Follow-up | 14
Not completed — Withdrawal by Subject | 36
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Idebenone
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (13.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 107
Region of Enrollment [Number; unit: participants]
  Netherlands | 8
  Austria | 6
  Belgium | 10
  France | 13
  Germany | 143
  United Kingdom | 20

OUTCOME MEASURES:

1. Primary Outcome: Measures of Safety and Tolerability: Nature and Frequency of Adverse Events (AEs)
Description: Global Overvbiew of accurance of AEs-Safety population. The Safety population included all subjects who received at least one dose of the study medication.
Time Frame: overall study, up to 24 months
Measure: Number; unit: participants
Arm/Group | Idebenone
Number analyzed (Participants) | 200
participants
  With at least one AE | 188
  With at least one drug-related AE | 109
  With at least one severe AE | 8
  With any significant AE | 54
  Death | 1
  Other serious adverse events than death | 48
  AEs leading to discontinuation | 26

2. Primary Outcome: Absolute Change in The International Cooperative Ataxia Rating Scale (ICARS)
Description: The International Cooperative Ataxia Rating Scale (ICARS) is a commonly used evaluation and is composed of four clinical sub-scores involving the following: posture and gait, limb coordination, speech and oculomotor function.The ICARS score is the total sum of the sub scores and ranges from 0 to 100, with 100 indicative of the most severely affected outcome.
Time Frame: Baseline, Month 12 and month 24
Population: Changes in Total ICARS Score for all patients completing the study (CC Population)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Idebenone
Number analyzed (Participants) | 139
units on a scale
  From Baseline to Month 12 | 1.41 (7.14)
  From Baseline to Month 24 | 2.88 (7.57)

3. Other Pre Specified Outcome: Measures of Safety and Tolerability: Physical Examinations and Vital Signs
Description: Assessment of the head, eyes, ears, nose, throat, heart, chest, lungs, abdomen, extremities, peripheral pulses, skin and any other physical conditions of note.
Time Frame: Month 1, 3, 6, 12, 18 and 24
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Measures of Safety and Tolerability: Electrocardiograms (ECGs)
Description: 12-lead ECG recordings were performed at every visit. Each ECG was measured using 3 complexes: PR interval in lead II or V2, QRS and QT intervals and heart rate in lead II, corrected QT intervals QTcB and QTcF.
Time Frame: Month 1, 3, 6, 12, 18 and 24
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Measures of Safety and Tolerability: Haematological and Biochemical Laboratory Parameters
Description: Safety haematological analysis were done at every visit. Analyses included red blood cell count, haemoglobin, haematocrit, red cell indices, white blood cell count including differential, platelet count Safety biochemistry were done at every visit. Analyses included sodium, potassium, chloride, bicarbonate, urea, creatinine, calcium, inorganic phosphate, glucose, total bilirubin, total protein, albumin, aspartate amiotransferase (AST), alanine aminotransferase (ALT), alkaline phosphotase, Gamma GT, creatine kinase (CK)^, cholesterol, triglycerides, uric acid.
Time Frame: Month 1, 3, 6, 12, 18 and 24
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Idebenone
Serious Adverse Events (participants affected / at risk) | 49/200
Other Adverse Events (participants affected / at risk) | 188/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idebenone (N=200)
Atrial fibrillation (Cardiac disorders) | 3 (4)
Atrial flutter (Cardiac disorders) | 2 (2)
cardiac failure (Cardiac disorders) | 1 (1)
talipes (Congenital, familial and genetic disorders) | 1 (2)
abdominal pain lower (Gastrointestinal disorders) | 1 (1)
diarrhoea (Gastrointestinal disorders) | 2 (2)
asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
streptococcal infection (Infections and infestations) | 1 (1)
dental caries (Gastrointestinal disorders) | 1 (1)
tooth disorder (Gastrointestinal disorders) | 1 (1)
fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
gastroenteritis (Gastrointestinal disorders) | 2 (2)
spinal disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
deep vein thrombosis (Vascular disorders) | 1 (1)
pulmonary embolism (Vascular disorders) | 1 (1)
ankle fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Humerus fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
lower respiratory tract infection (Infections and infestations) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Reflux oesophagitis (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Pelvic fracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1)
influenza (Infections and infestations) | 1 (1)
fibula fracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Tibia fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
proctitis (Gastrointestinal disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2)
femur fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
myocardial infarction (Cardiac disorders) | 1 (1)
abdominal pain upper (Gastrointestinal disorders) | 1 (1)
calculus ureteric (Renal and urinary disorders) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 1 (1)
epilepsy (Nervous system disorders) | 1 (1)
torticollis (Musculoskeletal and connective tissue disorders) | 1 (1)
salmonella sepsis (Infections and infestations) | 1 (1)
scoliosis (Musculoskeletal and connective tissue disorders) | 2 (2)
prostatitis (Reproductive system and breast disorders) | 1 (1)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
radiculopathy (Nervous system disorders) | 1 (1)
thyroid cancer (Endocrine disorders) | 1 (1)
paraplegia (Nervous system disorders) | 1 (1)
hand fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
wrist fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
corneal erosion (Eye disorders) | 1 (1)
ventricular tachycardia (Cardiac disorders) | 1 (1)
hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
liver injury (Injury, poisoning and procedural complications) | 1 (1)
fall (Injury, poisoning and procedural complications) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idebenone (N=200)
abdominal pain upper (Gastrointestinal disorders) | 16 (16)
diarrhoea (Gastrointestinal disorders) | 37 (37)
nausea (Gastrointestinal disorders) | 20 (20)
vomiting (Gastrointestinal disorders) | 11 (11)
pyrexia (General disorders) | 10 (10)
bronchitis (Infections and infestations) | 12 (12)
cystitis (Infections and infestations) | 12 (12)
influenza (Infections and infestations) | 19 (19)
nasopharyngitis (Infections and infestations) | 67 (67)
fall (Injury, poisoning and procedural complications) | 13 (13)
back pain (Musculoskeletal and connective tissue disorders) | 17 (17)
pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (15)
dizziness (Nervous system disorders) | 10 (10)
headache (Nervous system disorders) | 52 (52)
depression (Psychiatric disorders) | 10 (10)
cough (Respiratory, thoracic and mediastinal disorders) | 19 (19)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No